CLINICAL TRIAL: NCT05293834
Title: Feasibility and Pilot Study of Virtual Reality Aggression Prevention Training (VRAPT) for (Forensic) Psychiatric Patients
Brief Title: Virtual Reality Aggression Prevention Training (VRAPT) for (Forensic) Psychiatric Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University Psychiatric Clinics Basel (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-02439; pk22Graf
Record Dates: First submitted 2022-01-24; First posted 2022-03-24 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Forensic Psychiatry
Keywords: Aggression Prevention; Virtual Reality; Virtual Reality Aggression Prevention Training (VRAPT)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VRAPT intervention group (Experimental): Data collection process:
  1. Pre-intervention (t0): patients self-reports and staff observation;
  2. VRAPT: 8-16 weeks;
  3. Post-intervention (t1): patients self-reports, staff observations, and qualitative interview with participants and VRAPT therapists conducted by research staff;
  4. Follow-up 12 weeks after completion of the intervention (t2): patients self-reports and staff observations.
  Interventions: Behavioral: Virtual Reality Aggression Prevention Training (VRAPT)

INTERVENTIONS:
Behavioral: Virtual Reality Aggression Prevention Training (VRAPT) — VRAPT consists of sixteen 45- to 60-minute sessions that take place once or twice per week (total duration of the intervention = 8 to 16 weeks). Session time and intensity will be adapted to the individual participant and the sessions will be delivered by specially trained VRAPT therapists in individual settings. The immersive and interactive three-dimensional virtual environment will be presented via headphones and head-mounted displays, using software developed by CleVR. In the virtual environment, participants will interact with virtual characters that are controlled by the psychotherapist and practice new skills . The therapy program is targeted at factors and processes related to aggression and the underlying theoretical framework is based on cognitive behavioural therapy and the General Aggression Model (GAM).
  The VRAPT consists of 4 phases:
  1. Introduction (Session 1)
  2. Inventory phase (Sessions 2-6)
  3. Skills-training (Sessions 6-15)
  4. Evaluation (Session 16)

SUMMARY:
Violent and aggressive behavior as well as disorders related to aggressive behavior are highly common in both adult and juvenile forensic psychiatric patients, and is also present in a subgroup of non-forensic psychiatric in- and out-patients. One promising new treatment option is Virtual Reality. A newly developed program in this area is the Virtual Reality Aggression Prevention Training (VRAPT). The purpose of the current feasibility and pilot study is to test VRAPT in a Swiss forensic and non-forensic psychiatric setting, including both adult and juvenile patients, and to examine whether VRAPT is an effective treatment method for aggressive behavior.

DETAILED DESCRIPTION:
Violent and aggressive behavior as well as disorders related to aggressive behavior are highly common in both adult and juvenile forensic psychiatric patients, and is also present in a subgroup of non-forensic psychiatric in- and out-patients. In order to minimize the risk for future violent offending it is important to intervene in these high-risk populations. Previous research showed that punishment alone is counterproductive for repeated offending behavior. In contrast, treatment was found to have a positive effect on reoffending (i.e., less reoffending). However, although knowledge about the treatment of (forensic) psychiatric patients has increased significantly in recent decades, it is still not fully understood what works for whom under which circumstances. One promising new treatment option is Virtual Reality. A newly developed program in this area is the Virtual Reality Aggression Prevention Training (VRAPT). This training is currently implemented and examined in correctional and forensic psychiatric facilities in the Netherlands and in Sweden. Results from the first randomized controlled trial (RCT) on the effectiveness of the intervention showed that the VRAPT group showed a decrease in some aggressive behaviors at post-test, but not anymore at 3-month follow-up. The purpose of the current feasibility and pilot study is to test VRAPT in a Swiss forensic and non-forensic psychiatric setting, including both adult and juvenile patients, and to gather information needed for the design of a large, international, high-quality, multicenter RCT. The research questions will address the effect of VRAPT on aggressive behavior, state-trait anger expression, stages of motivational change, emotion regulation, and therapeutic alliance. The present investigation will be the first study to include juvenile forensic psychiatric patients as well as to test VRAPT in Switzerland, thereby increasing the generalizability of the research to other populations. Furthermore, it will be the first time VRAPT will be tested in a non-forensic psychiatric sample exhibiting aggressive behaviour. In addition, it will address problem awareness and therapy motivation as possible factors influencing treatment outcome, and address some of the limitations of previous research.

ELIGIBILITY:
Inclusion Criteria:

* forensic and non-forensic psychiatric in- and out-patients of the Forensic Department or Adult Department of the Psychiatric University Hospitals Basel with aggressive behavior problems according to their clinical treatment team (which includes senior medical doctor, therapist, nursing staff).

Exclusion Criteria:

* insufficient German language skills (in speech or reading);
* intellectual disabilities (IQ < 70);
* epilepsy;
* acute psychotic state.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Aggression Questionnaire | At pre-intervention (t0), post-intervention (t1 = 8-16 weeks after VRAPT), and 12 weeks Follow-up (t2)
  To examine the effect of VRAPT on self-reported aggressive behavior in forensic and non-forensic psychiatric patients. The Aggression Questionnaire measures an individual's aggressive responses and the ability to channel those responses in a safe, constructive manner. It consists of 34 items, scored on the following scales: Physical Aggression, Verbal Aggression, Anger, Hostility, Indirect Aggression. The respondent rates each item on a 5-point scale ranging from "Not at all like me" to "Completely like me."
Change in Social Dysfunction and Aggression Scale (SDAS) | At pre-intervention (t0) and post-intervention (t1 = 8-16 weeks after VRAPT), and 12 weeks Follow-up (t2)
  To examine the effect of VRAPT on observed aggressive behavior in forensic and non-forensic psychiatric patients. The Social Dysfunction and Aggression Scale (SDAS) consists of 9 items (SDAS-9) covering outward aggression and 2 items (SDAS-2) covering inward aggression. It provides systematic recording of staff observations on a broad range of aggressive behaviour. Illustrative examples are: irritability, e.g., difficulty controlling reactions; negativism, e.g., not wanting to cooperate; directed verbal aggressiveness, e.g., insulting people personally. All 9 items are scored along a 4-point scale ranging from "Absent" to "Severely present".

SECONDARY OUTCOMES:
Change in state-trait anger expression | At pre-intervention (t0), post-intervention (t1 = 8-16 weeks after VRAPT), and 12 weeks Follow-up (t2)
  To examine how VRAPT affects the self-reported state-trait anger expression in forensic and non-forensic psychiatric patients using the State-Trait Anger Expression Inventory-2 (STAXI-2). The STAXI-2 is a psychological assessment tool designed to examine participants' experience, expression, and control of anger. Scores range from 0 to 80, with higher scores indicating higher levels of anger and worse emotional regulation.
Change in stages of change | At pre-intervention (t0), post-intervention (t1 = 8-16 weeks after VRAPT), and 12 weeks Follow-up (t2)
  To examine how VRAPT affects the self-reported stages of change in forensic and non-forensic psychiatric patients using an adapted version of the University of Rhode Island Change Assessment-Domestic Violence (URICA-DV). This tool helps helps clinicians understand an individual's motivation and readiness to alter their abusive behavior. Scores range from 8 to 40, with higher scores indicating a greater readiness to change behavior.
Change in emotion regulation | At pre-intervention (t0), post-intervention (t1 = 8-16 weeks after VRAPT), and 12 weeks Follow-up (t2)
  To examine how VRAPT affects the self-reported emotion regulation in forensic and non-forensic psychiatric patients using the Difficulties in Emotion Regulation Scale. This self-report questionnaire measures difficulties in areas such as emotional awareness, clarity, acceptance, impulse control, goal-directed behavior, and access to emotion regulation strategies. Responses are rated on a scale, typically ranging from 1 (almost never) to 5 (almost always), to evaluate the frequency and severity of these difficulties.
Assessment of VRAPT experience | At post-intervention (t1= 8-16 weeks after VRAPT)
  To examine how VRAPT is experienced by patients, the I-group Presence Questionnaire (IPQ) and the Virtual Reality Sickness Questionnaire (VRSQ) are used. The IPQ helps to determine how the sense of presence in the virtual reality environment affects the delivery and effect of VRAPT, while the VRSQ assess cybersickness. The IPQ, with scores ranging from 0 to 80, measures individuals' beliefs and perceptions about their illness, where higher scores indicate more negative or maladaptive beliefs. The VRSQ, with scores ranging from 0 to 120, assesses vulnerability in interpersonal relationships, with higher scores suggesting greater vulnerability and worse relational health.
Assessment of VRAPT acceptance | At post-intervention (t1= 8-16 weeks after VRAPT)
  To examine how VRAPT is accepted, interviews are conducted with patients and therapists.
Change in therapeutic alliance | At pre-intervention (t0), post-intervention (t1 = 8-16 weeks after VRAPT), and 12 weeks Follow-up (t2)
  To examine how the therapeutic alliance with non-forensic psychiatric patients develops through the course of VRAPT, the short revised version of the Working Alliance Inventory (WAI-SR) is used. This brief, self-report measure evaluates three key components of the quality of the therapeutic alliance between a patient and therapist: bond, task agreement, and goal agreement. The responses are rated on a scale, typically ranging from 1 (seldom) to 7 (always), to capture the strength and effectiveness of the therapeutic relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Cyril Boonmann, PhD, Principal Investigator — Psychiatric University Hospitals (UPK) Basel
Locations (1):
- Psychiatric University Hospitals (UPK) Basel, Basel, Canton of Basel-City, Switzerland